CLINICAL TRIAL: NCT02589158
Title: Steady-state Pharmacokinetics of Atazanavir/Cobicistat and Darunavir/Cobicistat Once Daily Over 72 Hours in Healthy Volunteers
Brief Title: SSAT067 PK of Atazanavir/Cobicistat and Darunavir/Cobicistat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT067
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: HIV
MeSH Terms: interventions — Atazanavir Sulfate; Cobicistat; cobicistat mixture with darunavir

ARMS (1):
- Evotaz®, washout, then Rezolsta® (Experimental): All participants will be administered Evotaz®) (atazanavir 300mg + cobicistat 150mg) once daily for 10 days, undergo a ten-day wash out period and then take Rezolsta® (darunavir 800mg + cobicistat 150mg) once daily for 10 days.
  Interventions: Drug: Evotaz; Drug: Rezolsta

INTERVENTIONS:
Drug: Evotaz — All participants will be administered Evotaz®) (atazanavir 300mg + cobicistat 150mg) once daily for 10 days
  Other Names: atazanavir and cobicistat
Drug: Rezolsta — All participants will be administered Rezolsta® (darunavir 800mg + cobicistat 150mg) once daily for 10 days.
  Other Names: darunavir and cobicistat

SUMMARY:
The purpose of this study is to look at the levels of three HIV medications: atazanavir, darunavir and cobicistat in the blood after drug intake has been stopped, in order to understand how long these drugs persist in the blood. The study will specifically look at blood levels of these three drugs after taking them every day for 10 days. Participants will take Evotaz (atazanavir and cobicistat) on a first stage and Rezolsta (darunavir and cobicistat) on a second stage.

If the participants decide to take part, the duration of the study will be up to 33 days plus a screening visit which will take place up to 28 days prior to the start of the study, and a follow up visit, which takes place 7 to 14 days after the last dose of study medication. This study is not randomised which means that all participants will receive all study medications in the same order.

The participant and the study doctor will know which study medications the participant is taking at all times during the study.

DETAILED DESCRIPTION:
Protocol Number: SSAT067

EudraCT Number: 2015-002956-28

Name of Investigational Product: Evotaz®, Rezolsta®

Name of active ingredients: Atazanavir, darunavir and cobicistat

Study title: Steady-state Pharmacokinetics of Atazanavir/Cobicistat and Darunavir/Cobicistat Once Daily Over 72 Hours in Healthy Volunteers

Phase of study: Phase I

Objectives:

Primary:

-To assess the steady-state pharmacokinetics of atazanavir/cobicistat and darunavir/cobicistat over 72 hours, in HIV negative healthy volunteers.

Secondary:

* To assess the inter subject variability in atazanavir, darunavir and cobicistat plasma concentrations over 72 hours
* To assess the safety and tolerability of atazanavir/cobicistat and darunavir/cobicistat over 10 days of administration to healthy volunteers
* To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure

Study design: 33 days (excluding screening and follow up), open label, pharmacokinetic study.

Indication: Not applicable

Methodology: Measurements of steady state pharmacokinetic profiles of plasma atazanavir/cobicistat and darunavir/cobicistat in male and female healthy volunteers.

Planned sample size: Up to 30 male and female healthy volunteers will be enrolled at baseline in order to achieve 16 completing the study

Summary of eligibility criteria: Healthy participants as determined by medical history, physical examination, 12-lead electrocardiogram, and clinical laboratory evaluations will be eligible to participate in the study. Women of childbearing potential must not be nursing or pregnant. Women of childbearing potential must have a negative pregnancy test at screening.

Number of study centres: One

Duration of treatment: 33 days (excluding screening and follow up visits)

Dose and route of administration: All participants will be administered Evotaz®) (atazanavir 300mg + cobicistat 150mg) once daily for 10 days, undergo a ten-day wash out period and then take Rezolsta® (darunavir 800mg + cobicistat 150mg) once daily for 10 days.

Criteria for evaluation:

* Pharmacokinetic parameters of atazanavir/cobicistat will be evaluated on blood drawn on day 10 at 0 (pre-dose), 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hours post dose and days 11 to 13 (up to 72 hours post dose).
* Pharmacokinetic parameters of darunavir/cobicistat will be evaluated on blood drawn on day 30 at 0 (pre-dose), 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24 hours post dose and days 31 to 33 (up to 72 hours post dose).
* Safety and tolerability of medications will also be assessed by questions, physical examination and laboratory parameters. These will be performed at regular intervals during the drug study.

Primary Endpoint:

-Steady state plasma concentrations of atazanavir/cobicistat and darunavir/cobicistat up to 72 hours post-dose.

Secondary End point:

* Safety and tolerability of the studied drugs over 10 days of administration.
* Relationship between genetic polymorphisms and exposure to the studied drugs.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive
5. ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
6. Women of childbearing potential (WOCBP - definition in Appendix 5) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 4 weeks after the study

   A female may be eligible to enter and participate in the study if she:
   1. is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
   2. is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:

      * Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 4 weeks after discontinuation of all study medications;
      * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
      * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see protocol appendix 5 for an example listing of approved IUDs);
      * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
      * Approved hormonal contraception (see protocol appendix 5 for a listing of examples of approved hormonal contraception) plus male condom;
      * Any other method with published data showing that the expected failure rate is <1% per year.
      * Any contraception method must be used consistently, in accordance with the approved product label and for at least 4 weeks after discontinuation of IP.
7. Men who have partners who are women of childbearing potential (WOCBP - definition in Appendix 5) must be using an adequate method of contraception to avoid pregnancy in their partner throughout the study and for a period of at least 4 weeks after the study (see inclusion criteria 6)
8. Willing to consent to their personal details being entered onto the TOPS database
9. Willing to provide proof of identity by photographic ID at screen and any subsequent visit
10. Registered with a GP in the UK

Exclusion Criteria:

1. Any clinically significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B surface antigen or C antibody
4. Positive blood screen for HIV-1 or 2 by antibody/antigen assay
5. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
6. History or presence of allergy to darunavir, atazanavir cobicistat or excipients (sodium methyl parahydroxybenzoate, lactulose, Hypromellose Colloidal silicon dioxide, Silicified microcrystalline cellulose Crospovidone, Magnesium stearate, Polyvinyl alcohol- partially hydrolysed, Macrogol 3350,Titanium dioxide, Talc, Iron oxide red, Iron oxide black, Lactose monohydrate, Magnesium stearate, Gelatine Yellow iron oxide, Indigocarmin (E132), White ink, Shellac,Titanium dioxide (E171), Ammonium hydroxide, Propylene glycol , Simethicone, Hypromellose, Polyvinyl alcohol- partially hydrolysed, Macrogol 3350)
7. Current or recent (within 3 months) gastrointestinal disease
8. Known intolerance of lactose monohydrate, sunset yellow aluminium lake (E110), and patients with galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
9. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
10. Exposure to any investigational drug (or placebo) or participation in a clinical study involving the donation of blood samples within 3 months of first dose of study drug
11. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
12. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 4 weeks after the end of the treatment period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To assess the steady-state pharmacokinetics of atazanavir/cobicistat and darunavir/cobicistat over 72 hours, in HIV negative healthy volunteers as measured by Ctrough | Days 10 and 30
  Trough concentration (Ctrough) is defined as the concentration at 24 hours after the observed drug dose
To assess the steady-state pharmacokinetics of atazanavir/cobicistat and darunavir/cobicistat over 72 hours, in HIV negative healthy volunteers, as measured by Cmax | Days 10 and 30
  Cmax defined as the maximum observed plasma concentration.
To assess the steady-state pharmacokinetics of atazanavir/cobicistat and darunavir/cobicistat over 72 hours, in HIV negative healthy volunteers, as measured by t1/2 | Days 10 and 30
  t1/2 = Elimination half-life
To assess the steady-state pharmacokinetics of atazanavir/cobicistat and darunavir/cobicistat over 72 hours, in HIV negative healthy volunteers, as measured by Tmax | Days 10 and 30
  Tmax = time point at Cmax
To assess the steady-state pharmacokinetics of atazanavir/cobicistat and darunavir/cobicistat over 72 hours, in HIV negative healthy volunteers, as measured by total drug exposure | Days 10 and 30
  Total drug exposure is expressed as the area under the plasma concentration-time curve from 0-24 hours after dosing (AUC0-24h) and 0-72 hours (AUC0-72h)

SECONDARY OUTCOMES:
To assess the inter subject variability in atazanavir, darunavir and cobicistat plasma concentrations over 72 hours | Days 10 and 30
To assess the safety and tolerability of the studied drugs over 10 days in HIV negative healthy volunteers, assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. | Screening (day -28) to follow-up visit (day 41-54)
To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by Peak plasma concentration (Cmax) | Day 1
To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by trough concentration (Ctrough) | Day 1
To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by Area under the plasma concentration versus time curve (AUC) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, Chelsea and Westminster Hospital NHS Foundation Trust, London, London, United Kingdom